CLINICAL TRIAL: NCT03729557
Title: Cardiovascular Remodeling in Living Kidney Donors With Reduced Glomerular Filtration Rate
Acronym: CENS
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Jon Arne Birkeland, Principal investigator, Medical doctor, PhD, Oslo University Hospital
Other Study IDs: 2016/1961
Record Dates: First submitted 2018-10-10; First posted 2018-11-02 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
Keywords: Kidney donor
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney Donors
  Interventions: Procedure: Nephrectomy
- Control group

INTERVENTIONS:
Procedure: Nephrectomy — Unilateral nephrectomy
  Groups: Kidney Donors

SUMMARY:
Chronic kidney disease (CKD) is highly frequent, and patients with advanced CKD are known to have a high risk of developing cardiovascular disease (CVD). However, little is known about the cardiovascular risk in patients with mildly reduced kidney function (reduced glomerular filtration rate, GFR), affecting up to 10% of the general population; and importantly, also affecting living kidney donors. Until recently it has been believed that donating a kidney does not represent any health hazard. However, a recent Norwegian epidemiological study suggested that kidney donors have an increased risk of CVD. The pathogenesis linking reduced kidney function to CVD is not known. Living kidney donors provide a unique model for investigating the mechanisms underlying increased risk of CVD in patients with reduced GFR because living kidney donors are healthy before donation. Thus, the main purpose of the Project is to investigate the mekanismes underlying the development of cardiovascular remodelling induced by a reduction in GFR.

ELIGIBILITY:
* Donor Group: persons selected as living kidney donors according to the Norwegian donor criteria and accepted for surgery at Rikshospitalet, Norway
* Control Group: persons fulfilling the criteria according to the Norwegian transplantation protocol for living kidney donors with one exeption: they do not have to be investigated with CT angiography which is not considered necessary.

Exclusion Criteria:

• Persons who do not meet the Norwegian donor criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The project is a prospective longitudinal parallel group study including persons selected as living kidney donors according to the Norwegian donor criteria and accepted for surgery at Rikshospitalet, Norway. The donors will be compared to a control group consisting of individuals evaluated for donation, but not found eligible and healthy family members related to donors. The control individuals will be age and sex matched to living kidney donors. Control individuals who accept to participate will go through the same test battery (the Norwegian transplantation protocol for living kidney donors) as living kidney donors and must fulfil these criteria before inclusion as controls.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass. | Before kidney donation (between one month and 1 day before surgery), new investigation 2,5, 5 and 10 years after kidney donation.
  Cardiac magnetic resonance imaging (CMRI) and echocardiography.
Change in left ventricular strain. | Before kidney donation (between one month and 1 day before surgery), new investigation 2,5, 5 and 10 years after kidney donation.
  CMRI and echocardiography.

SECONDARY OUTCOMES:
Change in arterial pulse wave velocity. | Before kidney donation (between one month and 1 day before surgery), new investigation 2,5, 5 and 10 years after kidney donation.
  CMRI
Change in intima and media thickness of aorta. | Before kidney donation (between one month and 1 day before surgery), new investigation 2,5, 5 and 10 years after kidney donation.
  CMRI Inflammation: biomarkers.
Change in the calsium/phosphate homeostasis. | Before kidney donation (between one month and 1 day before surgery), new investigation 2,5, 5 and 10 years after kidney donation.
  DXA-scan.
Change in inflammation-marker. | Before kidney donation (between one month and 1 day before surgery), new investigation 2,5, 5 and 10 years after kidney donation.
  Biomarker: high sensitive CRP

CONTACTS AND LOCATIONS:
Overall Officials: Jon Arne Birkeland, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brobak KM, Halvorsen LV, Aass HCD, Soraas CL, Aune A, Olsen E, Bergland OU, Rognstad S, Blom KB, Birkeland JAK, Hoieggen A, Larstorp ACK, Solbu MD. Novel biomarkers in patients with uncontrolled hypertension with and without kidney damage. Blood Press. 2024 Dec;33(1):2323980. doi: 10.1080/08037051.2024.2323980. Epub 2024 Apr 12. PMID 38606688
- [Derived] Blom KB, Bergo KK, Espe EKS, Rosseland V, Grotta OJ, Mjoen G, Asberg A, Bergan S, Sanner H, Bergersen TK, Bjornerheim R, Skauby M, Seljeflot I, Waldum-Grevbo B, Dahle DO, Sjaastad I, Birkeland JA. Cardiovascular rEmodelling in living kidNey donorS with reduced glomerular filtration rate: rationale and design of the CENS study. Blood Press. 2020 Apr;29(2):123-134. doi: 10.1080/08037051.2019.1684817. Epub 2019 Nov 13. PMID 31718316